CLINICAL TRIAL: NCT00207857
Title: Test-Retest Reliability of Pulmonary Function Tests in Patients With Duchenne's Muscular Dystrophy
Status: Withdrawn | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: Duchenne's Muscular Dystrophy
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Duchenne's Muscular Dystrophy; Scoliosis
Keywords: Duchenne's Muscular Dystrophy; Scoliosis
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Scoliosis

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- With and Without PFTs

SUMMARY:
Nearly all patients with Duchenne's Muscular Dystrophy (DMD) have scoliosis. Posterior instrumented spinal fusion, which is a surgery to correct scoliosis, has been shown to improve quality of life and satisfaction of both parents and families. The progressive muscular weakness leads to the development of scoliosis soon after the child has become unable to walk. The muscular weakness and scoliosis also affect the pulmonary function of these children. Pulmonary Function Tests (PFT) have been used to determine "pulmonary fitness" prior to surgery as a way to determine how well or if the child will tolerate surgery. Children with poor results on the PFT are determined to be too fragile to tolerate such a large operation. The physicians conducting this study feel that the PFT may be inaccurate and that this may not be the best single test to determine "pulmonary fitness". The physicians conducting the study think things like the time of day the study is done, how tired you are when you complete the test, and how well you understand the test may affect the results of the test.

DETAILED DESCRIPTION:
All patients with DMD have routine PFT's every six months as standard of care. You will be randomized in to one of two groups. The group assignment will be chosen by chance, similar to flipping a coin. If you are assigned to group one you will first have your regularly scheduled PFT in the morning. You will be asked to complete a second PFT that afternoon as least 4 hours after the first PFT. You will then be asked to come back to the clinic in two weeks and repeat these PFT's, once in the morning and once in the afternoon at least 4 hours apart. Each PFT will take approximately 10 to 15 minutes. If you are assigned to group two, you will have your regularly scheduled PFT in the morning and then a second test in the afternoon at least four hours after the first test. After the second PFT you will receive training from a Respiratory Therapist. You will receive teaching handouts to take home and an incentive spirometer and peak flow meter to practice with. You will be asked to practice these tests 2 times a day and record your results. You will then be asked to come back to the clinic in two weeks to repeat 2 PFT's, once in the morning and again at least 4 hours later. All participants will be asked how they feel at the time of testing.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Duchenne's Muscular Dystrophy with diagnosed confirmed by a neurologist
* No longer able to ambulate for any meaningful amount of time
* No previous spinal operation

Exclusion Criteria:

* Any other type of muscular dystrophy or spinal muscular atrophy
* Tracheotomy
* Contractures of the upper extremities that would preclude using arm span as an estimation for height
* Previous spinal surgery
* Asthma, recurrent pneumonia, or other chronic lung disease

Ages: 6 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2004-03; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Estimated)

PRIMARY OUTCOMES:
PFT training | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tim Schrader, MD, Principal Investigator — Children's Orthopaedics of Atlanta
Locations (1):
- Children's Healthcare of Atlanta @ Scottish Rite, Atlanta, Georgia, United States